CLINICAL TRIAL: NCT02625805
Title: Evaluation of the Ability for Monitoring Dynamics in ADD/ADHD With an Easy to Use EEG
Brief Title: Evaluation of Use of Brain Activity Monitoring Dynamics in ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brainmarc Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLD5
Record Dates: First submitted 2015-12-07; First posted 2015-12-09 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2016-07

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Participants diagnosed with ADD/ADHD (Experimental): EEG monitoring (MindWave by NeuroSky and EPOC by Emotiv) and Methylphenidate administration
  Interventions: Device: EEG monitoring (MindWave by NeuroSky); Device: EEG monitoring (EPOC by Emotiv); Drug: Methylphenidate
- Healthy participants (Experimental): EEG monitoring (MindWave by NeuroSky and EPOC by Emotiv) and Methylphenidate administration
  Interventions: Device: EEG monitoring (MindWave by NeuroSky); Device: EEG monitoring (EPOC by Emotiv); Drug: Methylphenidate

INTERVENTIONS:
Device: EEG monitoring (MindWave by NeuroSky) — EEG evaluation will be conducted for duration of 10 minutes. 5 minutes without auditory stimulation and 5 minutes with auditory stimulation performed using standard headphone or earphones to reduce external noises. Additional EEG monitoring will be performed during performance of a computerized test using MindWave Headset.
Device: EEG monitoring (EPOC by Emotiv) — EEG evaluation will be conducted for duration of 10 minutes. 5 minutes without auditory stimulation and 5 minutes with auditory stimulation performed using standard headphone or earphones to reduce external noises.
Drug: Methylphenidate — Methylphenidate will be administered to each of the study participants in both groups in one of the two days on the study selected randomly.

SUMMARY:
This study evaluates the ability to support diagnosis and monitor of the dynamics in ADD/ADHD subjects with an easy to use EEG Device.

DETAILED DESCRIPTION:
The study will be conducted in two arms (arm I and arm II). In arm I, participants diagnosed with ADD/ADHD. In arm II, healthy participants.

The status of the participants will be evaluated with questionnaires computerized test and EEG characteristics will be collected for all study participants. .

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 -45 years.
* Able and willing to comply with all study requirements.

Diagnosed with ADD/ADHD based on clinical evaluation based on the questionnaires:

* Adult ADHD Self-Report Scale (ASRS)
* Wender-Utah Rating Scale
* Positive And Negative Affect Schedule (PANAS)

Exclusion Criteria:

Diagnosed with Psychotic or bipolar disorder.

* Diagnosed with a substantial Neurological disorder or general medical condition with an effect on EEG patterns such as Epilepsy or stroke
* A user of recreational or illicit drugs or has had a recent history (six months) of drug or alcohol abuse or dependence.
* Cognitive impairment.
* Hearing disorder and/or known ear drum impairment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Measurements of brain electrical signal in Micro volt. | 2 weeks
  Measurements of brain electrical signal in Micro volt will be quantified by an algorithm and correlated to ADHD state as evaluated by participants questionnaires, and computerized test.

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Bloch, MD, Principal Investigator — Shalvata Hospital
Locations (1):
- Shalvata Hospital, Hod HaSharon, Israel